CLINICAL TRIAL: NCT06926387
Title: An Open-label, Randomized, Single-dose, Oral Administration, 2-sequence, 2- Period, Crossover Study to Evaluate Bioequivalence Between YHP2407 and YHR2502 in Healthy Subjects
Brief Title: Bioequivalence Study betweenYHP2407 and YHR2502 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP2407-101
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer
Keywords: Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A(RT) (Experimental): 20 subjects, Cross-over, Single dose YHR2502 on period
  1, Single dose of YHP2407 on period 2
  Interventions: Drug: YHP2407; Drug: YHR2502
- B(TR) (Experimental): 20 subjects, Cross-over, Single dose of YHP2407 on period 1, Single dose of YHR2502 on period 2
  Interventions: Drug: YHP2407; Drug: YHR2502

INTERVENTIONS:
Drug: YHP2407 — Test drug: YHP2407, Comparator: YHR2502
Drug: YHR2502 — Test drug: YHP2407, Comparator: YHR2502

SUMMARY:
A randomized, open-label, single-dose, 2-sequence, 2-period, crossover clinical trial to investigate the bioequivalence between YHP2407 and YHR2502 in healthy volunteers

DETAILED DESCRIPTION:
40 healthy subjects will be randomized to one of the 2 groups in the same ratio.

Subjects in group 1 will be administered "comparator" and "YHP2407" by crossover design on period 1, 2. Subjects in group 2 will be administered "YHP2407" and "comparator" by crossover design on period 1, 2.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30 kg/m2
* Those without clinically significant congenital or chronic diseases

Exclusion Criteria:

* Those who have participated in a bioequivalence study or other clinical trials and have been administered with investigational products in 6 months prior to the first administration.
* Others who are judged ineligible to participate in the trial by the principal investigator.
* Female volunteers who are pregnant, suspected to be pregnant or breastfeeding.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-6 hours
  Area under the plasma drug concentration-time curve [AUCt] of Cefaclor Hydrate
Maximum plasma concentration [Cmax] | 0-6 hours
  Maximum plasma concentration [Cmax] of Cefaclor Hydrate

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] | 0-6 hours
  Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] of Cefaclor Hydrate
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] | 0-6 hours
  Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] of Cefaclor Hydrate
Time of peak concentration [Tmax] | 0-6 hours
  Time of peak concentration [Tmax] of Cefaclor Hydrate
Terminal phase of half-life [t1/2] | 0-6 hours
  Terminal phase of half-life [t1/2] of Cefaclor Hydrate

CONTACTS AND LOCATIONS:
Overall Officials: Hyejin Lim, Principal Investigator — Gimpo Woori Hospital
Locations (1):
- Gimpo Woori Hospital, Gimpo-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No